CLINICAL TRIAL: NCT02041429
Title: Phase II Study of Combination Ruxolitinib (INCB018242) With Preoperative Chemotherapy for Triple Negative Inflammatory Breast Cancer Following Completion of a Phase I Combination Study in Recurrent/Metastatic Breast Cancer
Brief Title: Ruxolitinib W/ Preop Chemo For Triple Negative Inflammatory Brca
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Beth Overmoyer MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-494
Record Dates: First submitted 2014-01-11; First posted 2014-01-22 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Recurrent Breast Cancer; Metastatic Breast Cancer
Keywords: Recurrent Breast Cancer; Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ruxolitinib; Paclitaxel

STUDY DESIGN:
Intervention Model Description: The multi-arm nature of this study is due to the dose-escalation design.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg (Experimental): Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 10 mg orally twice daily for 4 cycles
  1 cycle = 21 days
  Participants with stable disease or better will have the opportunity to continue on single agent 10 mg Ruxolitinib until disease progression, unacceptable toxicity or patient withdrawal.
  Interventions: Drug: Ruxolitinib; Drug: Paclitaxel
- Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg (Experimental): Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 15 mg orally twice daily for 4 cycles
  1 cycle = 21 days
  Participants with stable disease or better will have the opportunity to continue on single agent 15 mg Ruxolitinib until disease progression, unacceptable toxicity or patient withdrawal.
  Interventions: Drug: Ruxolitinib; Drug: Paclitaxel
- Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg (Experimental): Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 20 mg orally twice daily for 4 cycles
  1 cycle = 21 days
  Participants with stable disease or better will have the opportunity to continue on single agent 20 mg Ruxolitinib until disease progression, unacceptable toxicity or patient withdrawal.
  Interventions: Drug: Ruxolitinib; Drug: Paclitaxel
- Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg (Experimental): Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 25 mg orally twice daily for 4 cycles
  1 cycle = 21 days
  Participants with stable disease or better will have the opportunity to continue on single agent 20 mg Ruxolitinib until disease progression, unacceptable toxicity or patient withdrawal.
  Interventions: Drug: Ruxolitinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Ruxolitinib
  Other Names: (INCB18424)
Drug: Paclitaxel
  Other Names: Taxol

SUMMARY:
This phase I/II research study is evaluating a combination of drugs called paclitaxel and ruxolitinib as a possible treatment for inflammatory breast cancer. Ruxolitinib is a newly discovered drug that has been shown to block a pathway (called the IL6/JAK/Stat pathway) that may be important in cancer, including breast cancer. Blocking this pathway may stop cancer cells from growing. Ruxolitinib has been approved by the FDA for patients with bone marrow disease, and this is the first study using this drug in combination with paclitaxel for breast cancer. Paclitaxel (also called Taxol) is an FDA drug approved for breast cancer patients. Paclitaxel works by blocking the small microtubules inside cancer cells and preventing cell growth. Information from laboratory experiments suggests that ruxolitinib might also have effects on breast cancer.These studies have shown that ruxolitinib may make paclitaxel more effective.

DETAILED DESCRIPTION:
This study has two phases. The objective of Phase I to find the maximum dose (MTD) of Ruxolitinib when combined with standard dose of paclitaxel given weekly for advanced or metastatic breast cancer. Three participants will be entered at a dose ruxolitinib equaling 10 mg orally twice daily with weekly paclitaxel. If no dose-limiting toxicity is seen after 6 weeks of treatment (two cycles), then the dose of ruxolitinib will be escalated using a standard 3+3 design, until 2 participants experience dose limiting toxicity (DLT). The dose below the DLT is designated the MTD and this dose of ruxolitinib will be used in the phase II preoperative study for triple negative IBC.

During Cycle 1 the participant will come into clinic every week. At each visit, the participant will have a physical exam and will be asked questions regarding general health and specific questions about any problems that the participant might be having with any medications. About 2-3 additional tablespoons of blood will be taken before the participant's begins ruxolitinib, on Cycle 2 Day 1, Cycle 3 Day 1, and at the end of the study for research blood tests. Because these tests are being performed for research, and their clinical usefulness is unknown, the participant will not receive the results of these tests. The investigator will assess the participant's tumor by CT scans or MRI every 2 cycles. In addition, if the participant has tumors that are visible or can be palpated (felt), then they will be measured by the participant's study doctor in the clinic. If the participant has had a history of cancer in the bones or suspected cancer in the bones, then a bone scan will be performed before the participant can begin ruxolitinib. The bone scan may be repeated every 2 cycles and at the end of the study if the participant study doctor believes it is clinically needed. Otherwise, it does not need to be repeated. Photographs may be taken of the participant's tumor to assess the tumor response to the treatment.

The phase II period of the study will treat triple negative inflammatory breast cancer participants with ruxolitinib combined with 12 weeks of weekly paclitaxel followed by standard care Doxorubicin and Cyclophosphamide (AC) chemotherapy, eligible participants will proceed to surgical mastectomy followed by radiation. The phase II study will begin once the phase I study has been completed.

During the phase II study, participants will have a research biopsy of the breast followed by one week of ruxolitinib given twice daily. A second research biopsy of the breast is then performed and the participants will then receive combination ruxolitinib (at the MTD dose defined in the phase I study) and standard dose paclitaxel for 12 weeks. Participants will be seen weekly during treatment. One week after completing the combination therapy, participants will receive standard dose doxorubicin and cyclophosphamide (AC) every 2 weeks for 4 cycles.

We will evaluate the effect of JAK inhibition by ruxolitinib on the tumor by comparing pSTAT3+ expression of the pre-treatment research biopsy with the pSTAT3+ expression on the second research biopsy performed after one week of ruxolitinib. Participants who have disease regression following 12 weeks of ruxolitinib and paclitaxel followed by AC chemotherapy will undergo mastectomy, and the amount of residual breast cancer will be assessed. We will correlate the degree of residual cancer in the mastectomy with the amount of pSTAT3+ expression seen in the research biopsies. We will be checking standard blood tests, IL-6 and CRP levels throughout the treatment to see if the levels change in response to ruxolitinib treatment. This may be an easier method of determining treatment efficacy. Standard radiation therapy will be given following mastectomy.

ELIGIBILITY:
Inclusion Criteria:

Phase I

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participants must have histologically confirmed breast cancer that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients may not have received > 2 prior chemotherapies for advanced disease.
* Either measurable or evaluable disease is allowed.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of ruxolitinib in participants <18 years of age, children are excluded from this study.
* Life expectancy of greater than 3 months.
* ECOG performance status ≤ 2 (see Appendix A).
* Participants must have normal organ and marrow function as defined below:
* Leukocytes ≥3,000/mcL
* Absolute neutrophil count ≥1,500/mcL
* Platelets ≥100,000/mcL
* Total bilirubin within normal institutional limits
* AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits or creatinine clearance ≥ 60 mL/min/1.73 m2 for subjects with creatinine levels about institutional normal
* Both men and women are allowed.
* The effects of ruxolitinib on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Phase I

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Participants may not be receiving any other study agents within 2 weeks of initiating treatment.
* Participants with untreated or uncontrolled brain metastases are excluded from this clinical trial. Patients with treated and stable (> 4 weeks) brain metastasis are allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib.
* Participants receiving any medications or substances that are strong inhibitors of CYP3A4 are ineligible. (Please refer to Appendix B for list and washout periods).
* Chronic corticosteroid use in excess of the equivalent of prednisone 10 mg once daily.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ruxolitinib is a JAK inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with ruxolitinib, breastfeeding should be discontinued if the mother is treated with ruxolitinib. These potential risks may also apply to other agents used in this study.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Clinically significant malabsorption syndrome.
* Prior chemotherapy or radiation administered within 2 weeks from initiating study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Overmoyer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lynce F, Williams JT, Regan MM, Bunnell CA, Freedman RA, Tolaney SM, Chen WY, Mayer EL, Partridge AH, Winer EP, Overmoyer B. Phase I study of JAK1/2 inhibitor ruxolitinib with weekly paclitaxel for the treatment of HER2-negative metastatic breast cancer. Cancer Chemother Pharmacol. 2021 May;87(5):673-679. doi: 10.1007/s00280-021-04245-x. Epub 2021 Feb 14. PMID 33585999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants registered from February 3rd 2014 to July 7th 2015
Pre-assignment Details: One participant who enrolled and never received treatment was excluded from further analyses.
Period: Overall Study
Arm/Group | Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg | Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg | Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg | Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg
Started | 3 | 4 | 7 | 6
Treated | 3 | 3 | 7 | 6
Evaluable for Dose Limiting Toxicity | 3 | 3 | 6 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 7 | 6
Not completed — Progressive Disease | 2 | 2 | 3 | 2
Not completed — Toxicity | 0 | 1 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — On Maintenance Therapy | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The analysis population represents all treated participants.
Groups:
- Phase I Dose Level 0:: Paclitaxel + Ruxolitiniib 10 mg Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 10 mg orally twice daily for 4 cycles
  1 cycle = 21 days
  Participants with stable disease or better will have the opportunity to continue on single agent 10 mg Ruxolitinib until disease progression, unacceptable toxicity or patient withdrawal.
- Phase I Dose Level 1:: Paclitaxel + Ruxolitiniib 15 mg Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 10 mg orally twice daily for 4 cycles
  1 cycle = 21 days
  Participants with stable disease or better will have the opportunity to continue on single agent 10 mg Ruxolitinib until disease progression, unacceptable toxicity or patient withdrawal.
- Phase I Dose Level 2:: Paclitaxel + Ruxolitiniib 20 mg Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 10 mg orally twice daily for 4 cycles
  1 cycle = 21 days
  Participants with stable disease or better will have the opportunity to continue on single agent 10 mg Ruxolitinib until disease progression, unacceptable toxicity or patient withdrawal.
- Phase I Dose Level 3:: Paclitaxel + Ruxolitiniib 25 mg Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 10 mg orally twice daily for 4 cycles
  1 cycle = 21 days
  Participants with stable disease or better will have the opportunity to continue on single agent 10 mg Ruxolitinib until disease progression, unacceptable toxicity or patient withdrawal.
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 0: | Phase I Dose Level 1: | Phase I Dose Level 2: | Phase I Dose Level 3: | Total
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 19
Age, Continuous [Mean (Full Range); unit: years] | 53 [46 to 61] | 46.7 [45 to 50] | 56.1 [39 to 75] | 51 [33 to 58] | 52.6 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 6 | 19
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 7 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 7 | 6 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 7 | 6 | 19
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants]
  00 Fully Active | 3 | 2 | 4 | 6 | 15
  01 Restricted | 0 | 1 | 3 | 0 | 4
Prior Lines of Chemotherapy for Metastatic Breast Cancer [Count of Participants; unit: Participants]
  Zero | 2 | 1 | 3 | 4 | 10
  One | 0 | 2 | 2 | 1 | 5
  Two | 0 | 0 | 1 | 1 | 2
  Three | 1 | 0 | 1 | 0 | 2
Received Prior Endocrine Therapy for Metastatic Breast Cancer [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 6 | 3 | 12
  No | 2 | 1 | 1 | 3 | 7
Received Prior Adjuvant Chemotherapy [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 5 | 5 | 14
  No | 0 | 2 | 2 | 1 | 5
Received Prior Adjuvant Endocrine Therapy [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 2 | 5 | 8
  No | 2 | 3 | 5 | 1 | 11
Estrogen and/or Progesterone Receptor Positive [Count of Participants; unit: Participants]
  Positive | 1 | 1 | 5 | 4 | 11
  Negative | 2 | 2 | 2 | 2 | 8
Triple Negative (Estrogen, Progesterone, Tyrosine-Protein Kinase erbB-2 receptors negative) [Count of Participants; unit: Participants]
  Triple Negative | 2 | 2 | 2 | 2 | 8
  Not Triple Negative | 1 | 1 | 5 | 4 | 11
Measurable Disease Present at Baseline [Count of Participants; unit: Participants]
  Total: Yes | 2 | 2 | 6 | 5 | 15
  Total: No | 1 | 1 | 1 | 1 | 4
  Visceral Disease: Yes | 3 | 3 | 2 | 4 | 12
  Visceral Disease: No | 0 | 0 | 5 | 2 | 7
  Disease in Breast / Lymph Nodes / Soft Tissue: Yes | 2 | 2 | 7 | 2 | 13
  Disease in Breast / Lymph Nodes / Soft Tissue: No | 1 | 1 | 0 | 4 | 6
  Bone Metastases: Yes | 1 | 1 | 4 | 3 | 9
  Bone Metastases: No | 2 | 2 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Ruxolitinib Maximum Tolerated Dose (MTD) [Phase I]
Description: Ruxolitinib MTD in combination with paclitaxel 80 mg/m2 intravenously (IV) weekly is determined by the number of patients who have dose limiting toxicity (DLT). See DLT primary outcome measure for definition
  * If a DLT was observed in 0 of 3 patients in a cohort, then 3 patients were enrolled to the next cohort using a 5mg higher dose of ruxolitinib.
  * If a DLT was observed in 1 of 3 patients in a cohort, then 3 additional patients were added, and then if no further DLTs were observed, 3 patients were enrolled to the next cohort using a 5mg higher dose of ruxolitinib.
  * The MTD is identified as the level BELOW the cohort where DLT occurred in less than one third of patients within the cohort.
  * If no DLT's are observed, the MTD is not reached.
Time Frame: Participants were assessed prior to each dose of paclitaxel with ruxolitinib; The observation period for MTD evaluation was the first 2 cycles of treatment. (Up to 8 weeks).
Population: The analysis population represents all evaluable for dose limiting toxicity participants.
Measure: Number; unit: mg
Groups:
- All Phase I Participants: Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib orally twice daily according to the established dose escalation schedule for 4 cycles
  1 cycle = 21 days Participants with stable disease or better will have the opportunity to continue on single agent Ruxolitinib at the established dose until disease progression, unacceptable toxicity or patient withdrawal.
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 18
mg | 15

2. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) [Phase I]
Description: DLT: (a) grade >2 non-hematologic, non-hepatic, organ toxicity not due to disease progression or another clearly identified cause except: alopecia of any grade; Grade 3 nausea, vomiting or diarrhea and grade 3 fasting hyperglycemia that resolves to grade<2 within 3 days and 7 days, respectively, with our without optimal medical management; and grade 3 fasting hyperglycemia within 3 days of glucocorticoid use; (b) grade >3 thrombocytopenia lasting more than 24 hours or associated with clinically significant bleeding; (c) grade >3 neutropenia lasting >4 days or accompanied with fever; (d) grade>3 anemia; grade>2 total bilirubin, aspartate and alanine aminotransaminase (AST and ALT), or alkaline phosphatase (ALP) lasting > 72 hours except: with baseline grade 2 as a result of liver metastases then levels (ALP, AST, ALT) >10x upper limit of normal is DLT; (e) delay in ability to administer paclitaxel more than 2 weeks due to toxicity.
Time Frame: Participants were assessed prior to each dose of paclitaxel with ruxolitinib; The observation period for DLT evaluation was the first 2 cycles of treatment. (Up to 8 weeks).
Population: The analysis population represents all treated participants. One patient in dose level 2 was replaced having gone off before completing 2 cycles due to progressive disease.
Measure: Number; unit: participants with DLT
Groups:
- Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg: Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 10 mg orally twice daily
  cycle duration=21 days
  Participants with stable disease or better after 4 cycles could continue with ruxolitinib alone.
- Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg: Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 15 mg orally twice daily
  cycle duration=21 days
  Participants with stable disease or better after 4 cycles could continue with ruxolitinib alone.
- Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg: Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 20 mg orally twice daily
  cycle duration=21 days
  Participants with stable disease or better after 4 cycles could continue with ruxolitinib alone.
- Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg: Paclitaxel 80 mg/m2 IV weekly + Ruxolitinib 25 mg orally twice daily
  cycle duration=21 days
  Participants with stable disease or better after 4 cycles could continue with ruxolitinib alone.
Arm/Group | Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg | Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg | Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg | Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg
Number analyzed (Participants) | 3 | 3 | 7 | 6
participants with DLT | 0 | 0 | 1 | 0

3. Secondary Outcome: Best Response [Phase I]
Description: Best Response on treatment was measured according Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. For target lesions, complete response (CR) is complete disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Progressive disease (PD) is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria. CR and PR required confirmation at 4 weeks (not less than 28 days).
Time Frame: Disease was evaluated radiologically every 2 cycles/6 weeks on treatment. Treatment duration was up to 9 months.
Population: The analysis population represents all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg | Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg | Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg | Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg
Number analyzed (Participants) | 3 | 3 | 7 | 6
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 1 | 0 | 0 | 3
  Stable Disease | 1 | 3 | 6 | 2
  Progressive Disease | 1 | 0 | 1 | 1

4. Secondary Outcome: All-Cause Neutropenia
Description: Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. All-grade neutropenia, a neutrophil deficiency, is determined using established methods.
Time Frame: Measured while on treatment and up to 30 days after coming off treatment. Up to 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg | Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg | Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg | Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg
Number analyzed (Participants) | 3 | 3 | 7 | 6
Participants | 2 | 1 | 5 | 3

5. Secondary Outcome: C-Reactive Protein Change From Baseline
Description: C-Reactive Protein biomarkers evaluated using established methods. Change in level after 2 cycles of therapy from baseline was measure.
Time Frame: From day 1 of cycle 1 to day 1 of cycle 3 (up to 8 weeks)
Population: Some participants did not have evaluable samples. 17 total participants provided samples.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg | Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg | Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg | Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg
Number analyzed (Participants) | 3 | 3 | 5 | 6
mg/L | -1.6 [-38.6 to 1.5] | -4.3 [-14.9 to 0] | -9.7 [-32.9 to -4.1] | 0.45 [-52.9 to 32.7]

6. Secondary Outcome: IL-6 Change From Baseline
Description: IL-6 biomarkers evaluated using established methods. Change in levels after 2 cycles of therapy from baseline was measure.
Time Frame: From day 1 of cycle 1 to day 1 of cycle 3 (up to 8 weeks)
Population: Some participants did not have evaluable samples. 17 total participants provided samples.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg | Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg | Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg | Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg
Number analyzed (Participants) | 3 | 3 | 5 | 6
pg/mL | 0 [0 to 21.7] | -0.2 [-2.6 to 0] | -2.7 [-13.4 to 2.6] | 0.6 [-14.1 to 33.3]

ADVERSE EVENTS:
Time Frame: Measured while on treatment and up to 30 days after coming off treatment. Up to 10 months
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg | Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg | Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg | Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 5/7 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 6/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg (N=3) | Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg (N=4) | Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg (N=7) | Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg (N=6)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 5 | 3
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 0: Paclitaxel + Ruxolitiniib 10 mg (N=3) | Phase I Dose Level 1: Paclitaxel + Ruxolitiniib 15 mg (N=4) | Phase I Dose Level 2: Paclitaxel + Ruxolitiniib 20 mg (N=7) | Phase I Dose Level 3: Paclitaxel + Ruxolitiniib 25 mg (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 4
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Edema limbs (General disorders) | 2 | 1 | 0 | 2
Fatigue (General disorders) | 3 | 2 | 3 | 6
Flu like symptoms (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 2
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 1
Gum infection (Infections and infestations) | 0 | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 2 | 1 | 3 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Weight gain (Investigations) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1 | 2
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes